CLINICAL TRIAL: NCT05190965
Title: Comparison Between Findings in Optical Coherence Tomography Angiography and in Fluorescein Angiography in Patients With Diapetic Retinopathy
Brief Title: Optical Coherence Tomography Angiography and in Fluorescein Angiography in Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Reda Mohamed Mahmoud, E.r.mohamed, Assiut University
Other Study IDs: FFDR
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: OctA .FFA Findings in DR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: OCTAngiography .FFangiography — octa.ffa findings in pts with diapetic retinopathy

SUMMARY:
Diabetic retinopathy (DR) is the leading cause of decreased vision in working age people. Patients with DR can develop macular edema and proliferative retinopathy which are major causes of visual impairment [1]. The potential of OCTA regarding diagnosis and follow up of DR has been shown in previous studies [2-4]. At present fluorescein angiography (FA) represents the gold standard in the diagnosis and staging of DR [5]. With FA vascular lesions like micro aneurysms (MAs), the size of areas of non-perfusion and of the foveal avascular zone (FAZ) and retinal neovascularisations can be reliably identified [6]. Al-though the capabilities of FA are well known, its use also contains some risks related to the intravenous injection of the dye, which can cause nausea, vomiting and allergic re actions and even anaphylactic shock [7]. Besides that, it also requires time and trained personnel [8]. Image acquisition by OCTA in contrast is not as time consuming and can be performed without taking any risks. Additionally, it provides a 3 dimensional cross sectional view of the retinal and choroidal layers with micro meter depth resolution, providing depth selective information of the retinal vasculature. This facilitates accurate diagnosis and follow up of retinal vascular diseases since significant insights into both morphology and perfusion status can be obtained simultaneously. Although various artifacts appear in OCTA images, a qualitative assessment is mostly possible [9].Early changes to be seen in OCTA in patients with non-proliferative DR are vascular remodelling bordering the FAZ, vascular tortuosity, narrowing of capillary lumen and capillary dilatation. These changes cannot be seen in the same manner in FA [10].In this study we investigated the size of the FAZ and the count of MAs in patients with DR.

ELIGIBILITY:
Inclusion Criteria:

* All Pts with confirmed type 2 diabetes of at least 6 months. Best corrected visual Acuity of 6/60 or higher (using asnellen chart) in each eye

Exclusion Criteria:

* Dense media opacities interfere with image FFA as dense cataract . Previous TTT mainly retinal laser photocoagulation or intra vitreal injection. History of ocular disease as glaucoma and retinal vascular occlusion . Previous ocular surgery.

Ages: 45 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All included patients are planned to have FFA and OCTA en face 3x3mm
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Compare findings in OCTA.Ffa in DR | Baseline
  Number of microaneurysm.degree of ischemia.size of FAZ

REFERENCES:
- [Background] Klein R, Moss SE, Klein BE, Davis MD, DeMets DL. Wisconsin Epidemiologic Study of Diabetic Retinopathy. XII. Relationship of C-peptide and diabetic retinopathy. Diabetes. 1990 Nov;39(11):1445-50. doi: 10.2337/diab.39.11.1445. PMID 2121570
- [Background] Ghasemi Falavarjani K, Al-Sheikh M, Akil H, Sadda SR. Image artefacts in swept-source optical coherence tomography angiography. Br J Ophthalmol. 2017 May;101(5):564-568. doi: 10.1136/bjophthalmol-2016-309104. Epub 2016 Jul 20. PMID 27439739